CLINICAL TRIAL: NCT04411368
Title: Impact of Respiratory Virus in Critically Ill Patients With Acute Respiratory Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Jongmin Lee, Assistant professor, Seoul St. Mary's Hospital
Other Study IDs: ICU_RES_VIRUS
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Acute Respiratory Failure; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal aspirates, Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study to evaluate the clinical impact of respiratory virus in the patients with acute respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 19 years
* Written informed consent by the patient or legally authorized representative
* Critical illness consistent with acute respiratory failure, to be enrolled within 24 hours of presentation

Exclusion Criteria:

* No informed consent
* A patient who is judged to be unable to make a voluntary decision by understanding information about this research due to cognitive vulnerability

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with presentation to ICU with critical illness compatible with acute respiratory failrue.
  * Definition of acute respiratory failure: Patients who met one of following criteria
  1. SaO2 < 90% on room air
  2. SaO2 < 92% on > 6L/min of oxygen
  3. Respiratory rates > 30/min, or sign of respiratory distress
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of respiratory viral infections | within 24 hours after intensive care unit (ICU) admission
  Rate of respiratory viral infections in patients with acute respiratory failure

SECONDARY OUTCOMES:
ICU mortality rate | Through study completion, an average of 1 year
  Association between respiratory viral infections and death in ICU and risk factors of death in patients with ARF
Hospital mortality rate | Through study completion, an average of 1 year
  Association between respiratory viral infections and death in hospital and risk factors of death in patients with ARF

CONTACTS AND LOCATIONS:
Overall Officials: Jongmin Lee, Study Director — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea